CLINICAL TRIAL: NCT02268656
Title: Preducted Effect-site Concentration of Propofol for I-gel Insertion During Anesthesia Induction
Brief Title: Effect-site Concentration of Propofol for I-gel Insertion During Anesthesia Induction With a Single-dose Dexmedetomidine
Acronym: D-pofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, Assistant professor, Gachon University Gil Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GCIRB2014-153
Record Dates: First submitted 2014-10-09; First posted 2014-10-20 (Estimated); Results first posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Igel
MeSH Terms: conditions — Ige Responsiveness, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- concentration of propofol in male (Other): after infusion of dexmedetomidine dexmedetomidine 0.5 mcg/kgfor 2 min, infusion of propofol as using target controlled infusion pump. Effect site concentration would be changed as the response to i-gel insertion as up and down method in male
  Interventions: Drug: propofol concentration
- concentration of propofol in female (Other): after infusion of dexmedetomidine dexmedetomidine 0.5 mcg/kgfor 2 min, infusion of propofol as using target controlled infusion pump. Effect site concentration would be changed as the response to i-gel insertion as up and down method in female
  Interventions: Drug: propofol concentration

INTERVENTIONS:
Drug: propofol concentration — First subjects start from effect site concentraion of 5ug/ml propofol, after insertion of i-gel, determine the next subjects' effect site concentraion would be increae or decrease 0.5 ug/ml as up and down method
  Other Names: up and down method

SUMMARY:
Before anethetic induction, infuse dexmedetomidine 0.5 mcg/kg for 2 minutes and after injection of lidocaine 30 mg, propofol infusion by using target controlled infusion (TCI) pump. Effect site concentraion of propofol start from 5 and changes the concentration as previous response to i-gel insertion as up and down methods

DETAILED DESCRIPTION:
Before anethetic induction, infuse dexmedetomidine 0.5 mcg/kg for 2 minutes and after injection of lidocaine 30 mg, propofol infusion by using target controlled infusion (TCI) pump. Effect site concentraion of propofol start from 5 and changes the concentration as previous response to i-gel insertion as up and down methods. Failure of previous subjects are defined as difficulty to mouth open, severe nausea and couph and laryngeal spasm, and not loss of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS I-II, 20-60 yrs old

Exclusion Criteria:

* predicted difficulty airway, recent URI, BMI > 30kg/m2, reactive airway disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

REFERENCES:
- [Derived] Choi JJ, Kim JY, Lee D, Chang YJ, Cho NR, Kwak HJ. Male patients require higher optimal effect-site concentrations of propofol during i-gel insertion with dexmedetomidine 0.5 mug/kg. BMC Anesthesiol. 2016 Mar 22;16:20. doi: 10.1186/s12871-016-0186-1. PMID 27004426

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was no one who was excluded from the study before and after assignment to groups
Groups:
- Concentration of Propofol in Male: after infusion of dexmedetomidine dexmedetomidine 0.5 mcg/kgfor 2 min, infusion of propofol as using target controlled infusion pump. Effect site concentration would be changed as the response to i-gel insertion as up and down method in male
  propofol: First subjects start from effect site concentraion of 5ug/ml propofol, after insertion of i-gel, determine the next subjects' effect site concentraion would be increae or decrease 0.5 ug/ml as up and down method
- Concentraion of Propofol Infemale: after infusion of dexmedetomidine dexmedetomidine 0.5 mcg/kgfor 2 min, infusion of propofol as using target controlled infusion pump. Effect site concentration would be changed as the response to i-gel insertion as up and down method in female
  propofol: First subjects start from effect site concentraion of 5ug/ml propofol, after insertion of i-gel, determine the next subjects' effect site concentraion would be increae or decrease 0.5 ug/ml as up and down method
Period: Overall Study
Arm/Group | Concentration of Propofol in Male | Concentraion of Propofol Infemale
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Concentration in Male: after infusion of dexmedetomidine dexmedetomidine 0.5 mcg/kgfor 2 min, infusion of propofol as using target controlled infusion pump. Effect site concentration would be changed as the response to i-gel insertion as up and down method in male
  propofol: First subjects start from effect site concentraion of 5ug/ml propofol, after insertion of i-gel, determine the next subjects' effect site concentraion would be increae or decrease 0.5 ug/ml as up and down method
- Concentraion in Female: after infusion of dexmedetomidine dexmedetomidine 0.5 mcg/kgfor 2 min, infusion of propofol as using target controlled infusion pump. Effect site concentration would be changed as the response to i-gel insertion as up and down method in female
  propofol: First subjects start from effect site concentraion of 5ug/ml propofol, after insertion of i-gel, determine the next subjects' effect site concentraion would be increae or decrease 0.5 ug/ml as up and down method
- Total: Total of all reporting groups
Arm/Group | Concentration in Male | Concentraion in Female | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (11) | 35 (9) | 35 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 20 | 20
  Male | 20 | 0 | 20
Region of Enrollment [Number; unit: participants]
  South Korea | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Propofol
Description: effect site concentration of propofol
Time Frame: from i-gel insertion up to 5 min
Population: Patients who infused dexmedetomidine and propofol for anesthesia
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Concentration in Male | Concentraion in Female
Number analyzed (Participants) | 20 | 20
ug/ml | 5.46 (0.26) | 3.82 (0.34)

ADVERSE EVENTS:
Time Frame: During administration of study drugs approximately 5 minutes
Description: Adverse Events that were monitored for systematically were hypotension, hypertension, bradycardia, and other mild / serious adverse event including all cause of mortality
Arm/Group | Concentration in Male | Concentraion in Female
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concentration in Male (N=20) | Concentraion in Female (N=20)
bradycardia (General disorders) | 1 (1) | 0 (0)
hypertension (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No